CLINICAL TRIAL: NCT04585776
Title: An Exploratory Study Assessing Time in Target Glucose Range Using a New Titration Scheme of LY900014 and Insulin Degludec in Patients With Type 1 Diabetes
Brief Title: A Study of LY900014 and Insulin Degludec in Participants With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17601; I8B-MC-ITSZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Results first posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY900014 + Insulin Degludec (Experimental): LY900014 (100 units/milliliter (U/mL)) is a prandial insulin administered subcutaneously (SC) 0-2 minutes before meals. Insulin degludec (100 U/mL) is a basal insulin administered once daily SC. Participants received individually adjusted insulin doses during the 35-day titration period. The target glucose values were: fasting glucose 80-110 milligrams per deciliter (mg/dL), overnight glucose excursion (the difference between bedtime and prebreakfast glucose levels) < or = +/- 30 mg/dL, postprandial glucose peak <140 mg/dL or <20% increase from premeal level. Following the titration period, there was an 11-day maintenance period during which the doses were kept unchanged unless for safety reasons.
  Interventions: Drug: LY900014; Drug: Insulin Degludec

INTERVENTIONS:
Drug: LY900014 — Administered SC
Drug: Insulin Degludec — Administered SC

SUMMARY:
In this study, participants with type 1 diabetes (T1D) will take the study drug LY900014 and insulin degludec. The reason for this study is to evaluate the amount of time with glucose values within target range.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have type 1 diabetes and have been treated with insulin therapy for at least 1 year
* Participants must be using Continuous Glucose Monitoring (CGM) with total CGM use ≥ 2 months in the prior 6 months
* Participants must have been on the same type of short acting insulin (Humalog U-100, Novolog, Admelog, or Apidra) for at least 30 days prior to screening
* Participants must have been treated with long-acting insulin degludec U-100 for at least 30 days prior to screening

Exclusion Criteria:

* Participants must not have had more than 1 emergency room visit or hospitalization due to poor glucose control within 6 months before screening
* Participants must not have had more than 1 episode of severe hypoglycemia within the last 90 days prior to screening
* Participants must not be taking certain diabetes medications that are not allowed for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - HealthPartners Institute dba International Diabetes Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Bergenstal RM, Bode BW, Bhargava A, Wang Q, Knights AW, Chang AM. Assessing Time in Range with Postprandial Glucose-Focused Titration of Ultra Rapid Lispro (URLi) in People with Type 1 Diabetes. Diabetes Ther. 2023 Nov;14(11):1933-1945. doi: 10.1007/s13300-023-01476-4. Epub 2023 Sep 23. PMID 37740871
- See also: A Study of LY900014 and Insulin Degludec in Participants With Type 1 Diabetes. — https://trials.lillytrialguide.com/en-US/trial/32HuxMAefU6YDbyMk6SNjR

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY900014 + Insulin Degludec
Started | 31
Received Atleast 1 Dose of Study Drug | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY900014 + Insulin Degludec: LY900014 (100 U/mL) is a prandial insulin administered SC 0-2 minutes before meals. Insulin degludec (100 U/mL) is a basal insulin administered once daily SC. Participants received individually adjusted insulin doses during the 35-day titration period. The target glucose values were: fasting glucose 80-110 mg/dL, overnight glucose excursion (the difference between bedtime and prebreakfast glucose levels) < or = +/- 30 mg/dL, postprandial glucose peak <140 mg/dL or <20% increase from premeal level. Following the titration period, there was an 11-day maintenance period during which the doses were kept unchanged unless for safety reasons.
Arm/Group | LY900014 + Insulin Degludec
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.20 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time With Sensor Glucose Values Between 70 and 180 Milligrams Per Deciliter (mg/dL) With Continuous Glucose Monitoring (CGM)
Description: Percentage of Time with Sensor Glucose Values Between 70 and 180 mg/dL (both inclusive) with CGM.
Time Frame: Day 46
Population: All participants who received at least one dose of study drug and had post-baseline sensor glucose values.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | LY900014 + Insulin Degludec
Number analyzed (Participants) | 31
percentage of time
  Day-time | 71.57 (14.370)
  Night-time | 65.76 (19.846)
  24-Hour Period | 70.18 (14.589)

2. Secondary Outcome: Insulin to Carbohydrate Ratio (ICR)
Description: ICR was evaluated to estimate how many carbohydrates will be covered by one unit of insulin.
Time Frame: Day 46
Population: All participants who received at least one dose of study drug and had post-baseline ICR values.
Measure: Mean (Standard Deviation); unit: grams per insulin unit (g/U)
Arm/Group | LY900014 + Insulin Degludec
Number analyzed (Participants) | 31
grams per insulin unit (g/U)
  Breakfast: number analyzed (Participants) | 30
  Breakfast | 9.03 (3.490)
  Lunch | 9.07 (3.423)
  Dinner | 9.11 (3.529)
  Across meals | 9.05 (3.398)

3. Secondary Outcome: Ratio of Prandial Dose to Total Daily Dose (TDD) of Insulin
Description: Prandial:TDD ratio
Time Frame: Day 46
Population: All participants who received at least one dose of study drug and had post-baseline values for prandial and total daily insulin dose.
Measure: Mean (Standard Deviation); unit: percentage of insulin dose
Arm/Group | LY900014 + Insulin Degludec
Number analyzed (Participants) | 29
percentage of insulin dose | 52.06 (12.282)

4. Secondary Outcome: Product of Insulin to Carbohydrate Ratio and Total Daily Dose (ICR×TDD)
Description: ICR×TDD is determined to evaluate the relationship between insulin to carbohydrate ratio (g/U) and the total daily insulin dose (U/day).
Time Frame: Day 46
Population: All participants who received at least one dose of study drug and had post-baseline values for ICR and TDD.
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | LY900014 + Insulin Degludec
Number analyzed (Participants) | 29
g/day
  Breakfast | 411.1 (169.77)
  Lunch | 421.3 (184.18)
  Dinner | 427.6 (206.98)
  Across meals | 420.0 (183.52)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 53 days)
Description: All participants who received at least one dose of study drug.
Arm/Group | LY900014 + Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT04585776/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04585776/SAP_001.pdf